CLINICAL TRIAL: NCT07390422
Title: Duodenal Recellularization Via Electroporation Therapy for Suboptimally Controlled Type II Diabetes Mellitus and Steatotic Liver Disease (DRESS-1 Study)
Brief Title: Duodenal ReCET for Suboptimally Controlled Type II Diabetes Mellitus and Steatotic Liver Disease
Acronym: DRESS-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stephen KK Ng, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2025.876
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolic Syndrome (MetS)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic duodenal recellularization via electroporation therapy (ReCET) (Experimental): ReCET procedure entails the ablation of the duodenal mucosa with irreversible electroporation (IRE)
  Interventions: Procedure: ReCET treatment

INTERVENTIONS:
Procedure: ReCET treatment — The ReCET procedure utilizes the ReCET catheter to deliver non-thermal pulsed electric field to the duodenum to induce cell regeneration. The catheter is introduced to the duodenum through the mouth using a guide wire and the therapy is applied to treat the duodenum under endoscopic visualisation, starting from D4 and repeated proximally. Approximately 10-18 cm of axial length of the duodenum is treated.

SUMMARY:
This study is designed to evaluate the efficacy, safety, and mechanisms of ReCET procedure in patients with T2DM and its effect on MASLD.

DETAILED DESCRIPTION:
This is a prospective, single-arm feasibility study enrolling individuals with type 2 diabetes mellitus (T2DM) who have failed to achieve adequate glycemic control with oral glucose-lowering medications. Participants will undergo the ReCET procedure and liver biopsies both prior to and after the procedure to evaluate its effects on metabolically associated fatty liver disease (MAFLD). They will be followed for 12 months to assess the primary endpoint and for a total of 2 years. Participants are permitted to undergo a repeat ReCET procedure once if they initially respond but experience a recurrence of suboptimal diabetes management between 1 and 2 years after the procedure. They will be followed up for an additional year after the repeated procedure.

ELIGIBILITY:
Inclusion Criteria:

* Duration of T2DM < 10 years
* BMI 18.5-40kg/m2
* Failure to achieve adequate HbA1c reduction (7.5 - 11%) after at least 3 months stable dosage of oral glucose lowering drugs

Exclusion Criteria:

* Previous treatment with ReCET or similar procedure
* Previous GI surgery that could preclude the ability to perform ReCET, or acute gastric and duodenal pathology that increased the risk of ReCET
* Type 1 DM, DM secondary to specific disease or having any history of ketoacidosis
* Patients on insulin
* Fasting C-peptide level <0.5ug/L
* Any inflammatory disease of the gastrointestinal tract such as Crohn's disease
* Abnormal pathologies or conditions of the gastrointestinal tract, including duodenal polyps, ulcers or upper gastrointestinal bleeding conditions within 3 months of study
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/microliter or known coagulopathy
* Currently taking prescription antithrombotic therapy (e.g., anticoagulant or antiplatelet agent) within 10 days prior to study and/or there is a need or expected need to use during the study period
* Currently taking medications known to cause significant weight gain or weight loss (e.g. chemotherapeutics)
* Patients who have used non-steroidal analgesics and anti-inflammatory drugs (NSAID) and corticosteroids in the past 1 month
* Underlying uncontrolled endocrine problem that leads to obesity, including and not limited to hypothyroidism, Cushing syndrome and eating disorder.
* Patients with contra-indications to endoscopy
* Patients with cirrhosis due to causes other than MASLD
* Malignancy
* Diagnosis of autoimmune connective tissue disorder (e.g. lupus erythematosus, scleroderma)
* Pregnant or breast feeding
* ASA grade IV & V
* Mental or psychiatric disorder; Drug or alcohol addiction
* Other cases deemed by the examining physician as unsuitable for safe treatment
* Refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 24 months post-procedure
  Change in HbA1c (%) from baseline to Month 24
Improvement of MAFLD | 12 months post-procedure
  Proportion of subjects with improvement of liver steatosis and without worsening of fibrosis on liver histology

SECONDARY OUTCOMES:
Total body weight loss (%TBWL) | 24 months post-procedure
  Percent total body weight loss (%TBWL) from baseline to Month 24
Incidence of adverse events | within 30 days post-procedure
  Adverse events relating to endoscopic intervention, graded according to the Common Terminology Criteria for Adverse Events (CTCAE)
Body fat percentage | 24 months post-procedure
  Changes in body fat percentage - measured by bioelectrical impedance analysis from baseline to Month 24
Change in Quality of Life | 24 months post-procedure
  measured by 36-Item Short Form Survey (SF-36) questionnaire - (score 0:worst - 100:best) from baseline to Month 24
Faecal microbiome | 24 months post-procedure
  changes in faecal microbiome from baseline to Month 24
Changes in background glucose lowering medications | 24 months post-procedure
  Changes in glucose lowering medications from baseline to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ng, FRCSEd(Gen), Principal Investigator — Prince of Wales Hospital, the Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided